CLINICAL TRIAL: NCT06948396
Title: IdentiFy attRibutes Of uNcontrolled Severe asThma Patients trEateD With Tezepelumab: Italian Clinical Practice Study With the New bioloGic targEting TSLP
Brief Title: Observational Study on the Clinical Profile of Patients With Uncontrolled Severe Asthma Treated With Tezepelumab in Italy
Acronym: FRONTEDGE
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5180R00031
Record Dates: First submitted 2025-04-09; First posted 2025-04-29 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Asthma
Keywords: Asthma, uncontrolled severe asthma
MeSH Terms: conditions — Asthma | interventions — tezepelumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Severe uncontrolled asthma patients: Adolescent and adult patients with severe uncontrolled asthma treated with tezepelumab will be enrolled in the study. Patients can be enrolled if they received at least one dose of tezepelumab either within the sampling program or as per routine clinical practice between February 2024 and March 2025.
  Interventions: Biological: Tezepelumab

INTERVENTIONS:
Biological: Tezepelumab — Tezepelumab is indicated as an add-on maintenance treatment in adult and adolescent ≥12 years patients with severe uncontrolled asthma despite high-dose inhaled corticosteroids plus long-acting β-agonists

SUMMARY:
This observational study aims to collect data in clinical practice on the clinical profile of patients treated with Tezepelumab from Q1 2024 to Q1 2025 according to the approved and reimbursed indication in Italy

DETAILED DESCRIPTION:
There is a current need to gain information on the clinical profile of patients eligible for treatment with Tezepelumab according to the approved and reimbursed indication in Italy. Moreover, being Tezepelumab the latest approved biologic drug for severe asthma, it is important to better understand clinical response to treatment in patients with high severe asthma burden as: patients with allergic-eosinophilic phenotype; patients with low eosinophils level; patients affected by severe asthma associated with sinonasal disease; biologic-naïve patients, as well as bio-treated patients. The present observational study aims at filling the above-mentioned knowledge gaps in the study population in terms of clinical course, disease control and clinical remission, use of healthcare resources (treatments, visits, hospitalizations), lung functions, biomarkers, and sinonasal outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Adult and adolescent patients (age ≥12 years) at the Index Date (i.e., first administration of tezepelumab);
2. Patients with severe uncontrolled asthma (diagnosed according to clinician's judgment as per ERS-ATS or GINA guidelines) requiring a stable treatment of high doses of ICS and a long acting β2 agonist ± additional asthma controller;
3. Patients who received at least one injection of tezepelumab from February 2024 to March 2025 , according to Italian reimbursement indications;
4. Patients who signed the ICF and privacy form.
5. Patients with continuous enrolment in the data source for at least 12-months before the index date.
6. Patients with at least three months of continuous enrolment in the data source after the index date.

Exclusion Criteria:

1. Patients with hypersensitivity to the active ingredient or any of the excipients of Tezspire;
2. Patients who received any biologic drug for the treatment of asthma in a clinical trial at any time during the 12-months prior to the index date.
3. Patients who, during the observation period, participated in studies imposing a specific patient's management strategy, which does not correspond to the site's normal clinical practice.

Ages: 12 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adolescent and adult patients with severe uncontrolled asthma treated with at least one dose of tezepelumab between February 2024 and March 2025 will be enrolled in the study.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-09-10 (Actual); Primary Completion 2027-05-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Demographic and Clinic characterization | Basal
  To describe demographic and clinical characteristics of a population of patients with severe asthma who initiated treatment with tezepelumab
COMORBIDITIES AND RELEVANT MEDICAL HISTORY | Basal
  To describe the respiratory and non-respiratory related conditions in patients with severe asthma who initiated treatment with tezepelumab

SECONDARY OUTCOMES:
Exacerbation rate | Basal, 12 months, 24 months
  To describe the annualized asthma exacerbation rate in the 12-month period before (baseline period) and up to 12 and 24-months (follow-up period) after initiating treatment with tezepelumab in patients with severe asthma.
mOCS (maintenance Oral Corticosteroids) and ICS (Inhaled Corticosteroids) use | Basal, 12 months, 24 months
  To describe the mOCS and ICS daily dose in the 12-month period before (baseline period) and up to 12 and 24-months (+/- 2 months, follow-up period) after initiating treatment with tezepelumab in patients with severe asthma
ACT (Asthma Control Test) score | Basal, 12 months, 24 months
  To describe asthma control (ACT score) from last ACT score recorded before index date (within 12-month baseline period) and up to 12 and 24-months (+/- 2 months, follow-up period) after initiating treatment with tezepelumab in patients with severe asthma. ACT score range 1-25 - 25 means sympthoms under control
Asthma Control Questionnaire (ACQ) score | Basal, 12 months, 24 months
  To describe ACQ score from last score recorded before index date (within 12-month baseline period) and up to 12 and 24-months (+/- 2 months, follow-up period) after initiating treatment with tezepelumab in patients with severe asthma. ACQ score range 0-6. 6 means severely uncontrolled
Lung function FEV1 (L) | Basal, 12 months, 24 months
  To describe lung function through FEV1 (Forced Expiratory Volume in 1 Second) from last measurement before index date (within 12-month baseline period) and up to 12 and 24-months (+/- 2 months, follow-up period) after initiating treatment with tezepelumab in patients with severe asthma.
Lung function FVC (L) | Basal, 12 months, 24 months
  To describe lung function through FVC (Forced vital capacity) from last measurement before index date (within 12-month baseline period) and up to 12 and 24-months (+/- 2 months, follow-up period) after initiating treatment with tezepelumab in patients with severe asthma.
Lung function % predicted FVC | Basal, 12 months, 24 months
  To describe lung function through % predicted FVC (Forced vital capacity) from last measurement before index date (within 12-month baseline period) and up to 12 and 24-months (+/- 2 months, follow-up period) after initiating treatment with tezepelumab in patients with severe asthma.
Lung function % predicted FEV1 | Basal, 12 months, 24 months
  To describe lung function through % predicted FEV1 (Forced expiratory volume in 1 second) from last measurement before index date (within 12-month baseline period) and up to 12 and 24-months (+/- 2 months, follow-up period) after initiating treatment with tezepelumab in patients with severe asthma.
Biomarkers - BEC (blood eosinophils count) | Basal, 12 months, 24 months
  To describe BEC (cells/microL (cells/mm3)) in the 12-month period before (baseline period) and up to 12 and 24-months (+/- 2 months, follow-up period) after initiating treatment with tezepelumab in patients with severe asthma.
Biomarkers - FeNO (Fractional exhaled Nitric Oxide) | Basal, 12 months, 24 months
  To describe FeNO (ppb) in the 12-month period before (baseline period) and up to 12 and 24-months (+/- 2 months, follow-up period) after initiating treatment with tezepelumab in patients with severe asthma. FeNo range 0-99
Biomarkers - IgE (Immunoglobulin E) | Basal, 12 months, 24 months
  To describe blood IgE (IU/mL) in the 12-month period before (baseline period) and up to 12 and 24-months (+/- 2 months, follow-up period) after initiating treatment with tezepelumab in patients with severe asthma.
Treatments | Basal, 12 months, 24 months
  To describe treatment of asthma in 12-month period before (baseline period) and up to 12 and 24-months (+/- 2 months, follow-up period) after initiating treatment with tezepelumab in patients with severe asthma.
Clinical Remission | 12 months, 24 months
  To describe frequency and characteristics of patients achieving partial and complete clinical remission after 12 months and 24 months of treatment (+/- 2 months) [Severe Asthma Network in Italy (SANI) 2023 definition] [Canonica G et al, 2023].

OTHER OUTCOMES:
Demographics and clinic characterization_clinic remission | 12 months, 24 months
  To describe baseline demographics and clinical characteristics associated with clinical remission, frequency and characteristics of tezepelumab-treated patients achieving clinical remission after 12 and 24 months.
HCRU - number of specialistic visits for asthma | Basal, 12 months, 24 months
  To describe total number of specialist visits for asthma in the 12-month period before (baseline period) and up to 12 and 24-months (follow-up period) after initiating treatment with tezepelumab in patients with severe asthma.
HCRU - number of hospitalization | Basal, 12 months, 24 months
  To describe total number of hospitalization the 12-month period before (baseline period) and up to 12 and 24-months (follow-up period) after initiating treatment with tezepelumab in patients with severe asthma.
HCRU - number of ER visits | Basal, 12 months, 24 months
  To describe total number of ER visits in the 12-month period before (baseline period) and up to 12 and 24-months (follow-up period) after initiating treatment with tezepelumab in patients with severe asthma.
NP clinical outcomes - NPS (Nasal Polyp Score) | Basal, 12 months, 24 months
  To describe NPS (0-8) among severe asthma patients with comorbid CRSwNP during the baseline and follow-up period (12 and 24 months of treatment). NPS score: reduced score indicates improvement
NP clinical outcomes - Lund-Mackay (LMK) score | Basal, 12 months, 24 months
  To describe LMK (0-24) among severe asthma patients with comorbid CRSwNP during the baseline and follow-up period (12 and 24 months of treatment). LMK 24 means complete opacity of all sinuses
NP clinical outcomes - Visual Analogue Scale (VAS) | Basal, 12 months, 24 months
  To describe VAS (0-40) among severe asthma patients with comorbid CRSwNP during the baseline and follow-up period (12 and 24 months of treatment). VAS 40 means higher pain
NP clinical outcomes - 22-item Sino-Nasal Outcome Test (SNOT-22) | Basal, 12 months, 24 months
  To describe SNOT-22 (0-110) among severe asthma patients with comorbid CRSwNP during the baseline and follow-up period (12 and 24 months of treatment). Higher scores indicate greater rhinosinusitis-related health burden
NP clinical outcomes - NP surgeries | Basal, 12 months, 24 months
  To describe number of NP surgeries among severe asthma patients with comorbid CRSwNP during the baseline and follow-up period (12 and 24 months of treatment). Higher scores indicate greater rhinosinusitis-related health burden
Subgroups | Basal, 12 months, 24 months
  To describe clinical outcomes from the primary, secondary, and/or exploratory objectives in sub-groups of interest
Tezepelumab treatment | 12 months, 24 months
  To describe duration of therapy with tezepelumab, discontinuation, and reasons for discontinuation after initiating treatment with tezepelumab.

CONTACTS AND LOCATIONS:
Locations (30):
- Italy (30):
  - Research Site, Garbagnate Milanese, Milano
  - Research Site, Cittadella, Padova
  - Research Site, Montebelluna, TV
  - Research Site, Aosta
  - Research Site, Avellino
  - Research Site, Bari
  - Research Site, Bergamo
  - Research Site, Brescia
  - Research Site, Cagliari
  - Research Site, Catania
  - Research Site, Catanzaro
  - Research Site, Civitanova Marche
  - Research Site, Ferrara
  - Research Site, Foggia
  - Research Site, Genova
  - Research Site, Lamezia Terme
  - Research Site, Massa Carrara
  - Research Site, Milan
  - Research Site, Modena
  - Research Site, Napoli
  - Research Site, Orbassano (TO)
  - Research Site, Padua
  - Research Site, Reggio Calabria
  - Research Site, Reggio Emilia
  - Research Site, Roma
  - Research Site, Salerno
  - Research Site, Sassari
  - Research Site, Torino
  - Research Site, Tradate (VA)
  - Research Site, Verona

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/